CLINICAL TRIAL: NCT07216586
Title: Comparing Opioid Consumption Following Total Knee Arthroplasty With The Perioperative Administration of Zynrelef Versus Adductor Canal Block
Brief Title: Zynrelef Versus Adductor Canal Block
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Colin A. McNamara, Professor of Orthopaedic Surgery, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20250529
Record Dates: First submitted 2025-10-10; First posted 2025-10-14 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Knee Osteoarthritis; Arthritis Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — bupivacaine-meloxicam drug combination; Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Zynrelef (HTX-011) with application procedure (Experimental): Participants in this group will receive intraoperative analgesia via application of ZYNRELEF (HTX-011) directly into the periarticular tissues at the surgical site following prosthesis implantation and prior to capsule closure. The medication will be applied by the surgeon using sterile technique per manufacturer instructions, targeting the posterior capsule, medial and lateral gutters, and surrounding soft tissues.
  Interventions: Drug: ZYNRELEF 400Mg-12Mg Extended-Release Solution
- Adductor canal block (ACB) (Active Comparator): Participants in this group will receive a postoperative ultrasound-guided adductor canal block performed by a board-certified anesthesiologist or regional anesthesia-trained provider. The procedure will be conducted under sterile conditions while the patient remains under spinal anesthesia.
  Interventions: Procedure: Ultrasound-Guided Adductor Canal Block; Drug: Ropivacaine 0.5% Injectable Solution

INTERVENTIONS:
Drug: ZYNRELEF 400Mg-12Mg Extended-Release Solution — A single 14 mL dose of HTX-011 containing 400 mg bupivacaine and 12 mg meloxicam will be applied intraoperatively to the surgical site. This FDA-approved formulation is designed to provide sustained analgesia for up to 72 hours following total knee arthroplasty.
  Other Names: HTX-011
  Arms: Zynrelef (HTX-011) with application procedure
Procedure: Ultrasound-Guided Adductor Canal Block — A board-certified anesthesiologist or regional anesthesia-trained provider will perform an ultrasound-guided adductor canal block under sterile conditions while the patient remains under spinal anesthesia. A high-frequency linear ultrasound probe will be used to visualize the adductor canal and saphenous nerve.
  Arms: Adductor canal block (ACB)
Drug: Ropivacaine 0.5% Injectable Solution — A single injection of 30 mL of 0.5% ropivacaine will be administered into the adductor canal to provide postoperative analgesia. This dose is standard for adductor canal blocks and is intended to minimize motor blockade while providing effective pain control.
  Arms: Adductor canal block (ACB)

SUMMARY:
To compare postoperative MME consumption 72 hours after TKA in patients receiving intraoperative periarticular HTX-011 (Zynrelef) instillation versus adductor canal block.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age
* Patients undergoing primary, unilateral total knee arthroplasty
* Ability to provide informed consent

Exclusion Criteria:

* Individuals under the age of 18
* Pregnant women
* Prisoners
* Adults unable to consent
* American Society of Anesthesiologists Physical Status score greater than 3
* Patients taking any of the following medications before surgery:
* Long-acting opioids within 3 days
* Any opioids taken within 24 hours
* Bupivacaine HCL within 5 days
* Chronic opioid use or patients with known or suspected daily use of opioids for seven or more consecutive days within 6 months before their scheduled surgery
* Illicit drug use determined by social history
* Alcohol abuse determined by a CAGE Substance Abuse Screening Tool Score of at least two or greater
* Patients with a known hypersensitivity (e.g., anaphylactic reactions and serious skin reactions) to any local anesthetic agent of the amide-type, NSAIDs, or to any of the other components of ZYNRELEF
* Patients with a history of asthma, urticaria, or other allergic-type reactions after taking aspirin or other NSAIDs. Severe, sometimes fatal, anaphylactic reactions to NSAIDs have been reported in such patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Mean Milligram Morphine Equivalents (MME) | 12, 16, 20, 24, 48, and 72 hours after surgery
  Mean cumulative milligram morphine equivalents (MME) administered at 4, 8, 12, 16, 20, 24, 48, and 72 hours following total knee arthroplasty (TKA). Values will be compared between patients receiving Zynrelef and those receiving adductor canal block (ACB)

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) pain scores | 4 hours after surgery and 6 weeks
  Pain scores assessed 4 hours after surgery and at 6 weeks follow up using the Visual Analog Scale (VAS) for pain assessment consists of a line drawn in the form of a ruler, and numbers from 0 to 10 (with 0 as "no pain" and 10 as "unbearable pain"
Hospital length of stay measured in hours | 7 days
  Average hospital length of stay measured in hours
Knee range of motion | Within 48 hours of surgery, 6 weeks follow up
  Knee range of motion will be measured in degrees using a standardized goniometer or equivalent clinical tool. Assessments will be conducted postoperatively (within 48 hours of surgery) and at 6-week follow-up. Higher degrees indicate improved joint mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Colin A. McNamara, MD,MBA, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No